CLINICAL TRIAL: NCT05591144
Title: Investigating the Efficacy of Short-term Oral Prednisone Therapy on Acute Subjective Tinnitus
Brief Title: Short-term Oral Prednisone for Acute Subjective Tinnitus
Acronym: STOP-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STOP for AST
Record Dates: First submitted 2022-10-16; First posted 2022-10-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-05

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — Prednisone; Ginkgo biloba extract; Ginkgo Extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STOP group (Experimental): a 10mg/d tapering 14-day course of oral prednisone intervention (the initial dose: 1mg/kg/day, max 60mg/day) in combination with ginkgo biloba agent (120mg, three times/day)
  Interventions: Drug: Prednisone tablet; Drug: Ginkgo Biloba Extract
- placebol group (Placebo Comparator): Patients took oral standardized Ginkgo biloba extracts (120 mg daily) three times a day.
  Interventions: Drug: Ginkgo Biloba Extract

INTERVENTIONS:
Drug: Prednisone tablet — The dose selection of oral prednisone is the maximum daily dose based on weight for 4 days, followed by a taper every 2 days, with the maximum duration to 14 days.
  Other Names: prednisone
  Arms: STOP group
Drug: Ginkgo Biloba Extract — Ginkgo biloba extracts are traditional Chinese medicine, which can improve microcirculation and provide good ameliorating effects for the treatment of tinnitus
  Other Names: ginkgo biloba

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of oral steroids in the acute tinnitus population. Participants will receive appropriate dosages of short-term prednisone and/or oral Ginkgo Biloba tablets.

DETAILED DESCRIPTION:
Researchers will compare the intervention group and placebo-control group to see whether short-term systemic steroid therapy is effective for acute tinnitus.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old;
2. a primary complaint of frequent occurrences of subjective tinnitus lasting at least 5 minutes within the past 3 months ;
3. a definition of normal hearing in line with the World Report on Hearing (2021), of which the average value of hearing threshold at 500, 1000, 2000, 4000 Hz in better ear was less than 20 decibels;
4. a score of more than 16 points on the Tinnitus Handicap Inventory (THI), which indicates that the level of tinnitus exceeds mild severity;
5. a state of good general condition.

Exclusion Criteria:

1. had previous history of middle ear pathology, apparent history of noise exposure, noise trauma or head injury;
2. had received treatment for their current condition before the study;
3. taken oral steroids within 3 months before randomization;
4. had hearing implants;
5. had participated in other clinical trials and have not terminated the trials;
6. had a history of known corticosteroid contraindications (including osteoporosis, peptic ulcers, poorly controlled hypertension, diabetes, chronic liver or renal insufficiency, tumorous condition, alcohol abuse, pregnancy, or taking estrogen-containing oral contraceptive steroids);
7. auditory hallucinations or other conditions deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
tinnitus handicap inventory (THI) | two weeks from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
tinnitus handicap inventory (THI) | four weeks from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
tinnitus handicap inventory (THI) | twelve weeks from baseline
  The THI is a self-administered test, including 25 questions with grades four categories of tinnitus severity: slight corresponding to a score of 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.

SECONDARY OUTCOMES:
visual analog scale (VAS) | two weeks from baseline
  The subjective perception of tinnitus loudness will be evaluated using a Visual Analog Scale (VAS). Participants will be instructed to rate the perceived loudness of their tinnitus on a scale ranging from 0, indicating "no loudness," to 10, representing "maximum imaginable loudness." Higher scores on this scale will correspond to greater perceived loudness of tinnitus symptoms.
visual analog scale (VAS) | four weeks from baseline
  The subjective perception of tinnitus loudness will be evaluated using a Visual Analog Scale (VAS). Participants will be instructed to rate the perceived loudness of their tinnitus on a scale ranging from 0, indicating "no loudness," to 10, representing "maximum imaginable loudness." Higher scores on this scale will correspond to greater perceived loudness of tinnitus symptoms.
visual analog scale (VAS) | twelve weeks from baseline
  The subjective perception of tinnitus loudness will be evaluated using a Visual Analog Scale (VAS). Participants will be instructed to rate the perceived loudness of their tinnitus on a scale ranging from 0, indicating "no loudness," to 10, representing "maximum imaginable loudness." Higher scores on this scale will correspond to greater perceived loudness of tinnitus symptoms.
the Athens Insomnia Scale-8 (AIS-8) | two weeks from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
the Athens Insomnia Scale-8 (AIS-8) | four weeks from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).
the Athens Insomnia Scale-8 (AIS-8) | twelve weeks from baseline
  The AIS comprises eight items that commonly measure difficulties in falling asleep or maintaining sleep to quantify the presence of insomnia. The higher the AIS score, the lower the sleep quality and mental status. The AIS identifies three types of sleep disorders: no insomnia (score below 4), suspicious (4-6), and insomnia (score between 7-24).

CONTACTS AND LOCATIONS:
Overall Officials: Shan Sun, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No